CLINICAL TRIAL: NCT00209794
Title: The Impact of Intermittent Malaria Treatment Administered Through the EPI Scheme on Malaria Morbidity in Mozambican Children
Brief Title: IPTi in Mozambican Infants for Malaria Prevention
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TIM
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Sulfadoxine-Pyrimethamine (Fansidar)

SUMMARY:
To evaluate if intermittent preventive treatment in infants (IPTi) consisting of SP [Fansidar] given through the EPI scheme alongside routine immunisations at 3, 4 and 9 months of age reduces de incidence of clinical malaria up to 12 months of age

DETAILED DESCRIPTION:
The study is a randomised, double blind, placebo-controlled trial of the antimalarial drug sulphadoxine-pyrimethamine administered intermittently at 3, 4 and 9 months of age through the EPI scheme at the time of routine immunisations.

Children will be randomized into placebo and SP treatment groups by block randomization, and it is expected a similar age distribution and a similar number of children in each group.

Doses of sulphadoxine (25 mg/kg)-pyrimethamine (1.25 mg/kg) (SP) or placebo will be given by a health assistant according to bodyweight (a quarter of a tablet for those <5kg, a half for those 5-10 kg, and a whole tablet for children >10 kg). The tablets will be crashed and diluted with water for their administration.

ELIGIBILITY:
Inclusion Criteria:

* Children from study area
* Signed informed consent

Exclusion Criteria:

* History of drug allergies

Max Age: 3 Months | Sex: All
Age Groups: Child
Enrollment: 1498
Dates: Start 2002-09; Study Completion 2005-12

PRIMARY OUTCOMES:
Incidence of first or only malaria episodes in each study cohort by 12 months of age.

SECONDARY OUTCOMES:
Incidence of first or only malaria episodes by group up to 12 months of age as per protocol analysis.
Incidence of first or only malaria episodes by group up to 24 months of age.
Incidence of multiple malaria episodes up to 12 months of age.
Incidence of multiple malaria episodes up to 24 months of age.
Incidence of overall and severe anaemia up to 12 months of age.
Incidence of overall and severe anaemia up to 24 months of age.
Proportion of humoral and cellular immune responses against malaria at 12 months of age.
Total number of admissions and outpatient attendances up to 24 months of age.
Prevalence of P falciparum parasitaemia and overall and severe anaemia at 12 months of age.
Proportion of humoral responses and geometric mean antibody titres of polio, DTP and Hepatitis B at 5 months and of measles at 9 and 12 months
Incidence of side effects in each group up to 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Principal Investigator — Center for International Health, Hospital Clinic de Barcelona
Locations (1):
- Centro de Investigaçao em Saude da Manhiça, Manhiça, Maputo Province, Mozambique

REFERENCES:
- [Derived] Mayor A, Serra-Casas E, Sanz S, Aponte JJ, Macete E, Mandomando I, Puyol L, Berzosa P, Dobano C, Aide P, Sacarlal J, Benito A, Alonso P, Menendez C. Molecular markers of resistance to sulfadoxine-pyrimethamine during intermittent preventive treatment for malaria in Mozambican infants. J Infect Dis. 2008 Jun 15;197(12):1737-42. doi: 10.1086/588144. PMID 18419347
- See also: Related Info — http://www.manhica.org